CLINICAL TRIAL: NCT05173103
Title: Multicenter Retrospective Observational (Descriptive) Study of Second-line Therapies After Progression to CDK4/6i in Association With Hormone Therapy, in Patients With HR+/HER2- Advanced Breast Cancer (HERMIONE 13)
Brief Title: Retrospective Study of 2nd-line Therapies After CDK4/6i + Hormonal Therapy in HR+/HER2- Advanced Breast Cancer
Acronym: HERMIONE-13
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: HERMIONE 13
Record Dates: First submitted 2021-11-19; First posted 2021-12-29 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2023-12

CONDITIONS: Advanced Breast Cancer; Hormone Receptor Positive Breast Carcinoma; HER2-negative Breast Cancer
Keywords: advanced breast cancer; hormonal therapy; CDK 4/6 inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Description of the choices for second line treatment, in the normal clinical practice of the centers adhering to the Hermione Network, in patients affected by advanced HR+/HER2- breast cancer who progressed after CDK4/6i in association with hormonal therapy.

DETAILED DESCRIPTION:
Multicenter retrospective observational study, describing therapeutic choices as second-line treatment in patients with HR + / HER2- advanced breast cancer in a real world setting, in centers adhering to the Hermione Network.

The study involves the analysis of patients with HR + / HER2- advanced breast cancer treated in second line after initial treatment failure with aromatase inhibitor or Fulvestrant + CDK4 / 6i (Palbociclib, Ribociclib or Abemaciclib).

Data will be collected from 150 patients with at least one radiological re-evaluation of disease during 2nd-line treatment from 01 January 2016 until 31 December 2020.

List of collected information: Patients' characteristics (gender, age at diagnosis, menopausal state); Disease definition at diagnosis (stage, tumour histology, hormonal status); Surgery (date of surgery, type of surgical approach); Neo-adjuvant treatment; Adjuvant treatment; Date of first relapse (and time since the end of adjuvant therapy); Locations of metastases, Biopsy of metastases, Hormonal receptor status; First-line treatment, hormonal therapy, Best response, Cause of treatment end; Second-line treatment, Best response (radiological re-evaluation), Toxicity, Cause of treatment end.

Demographics, baseline characteristics (including tumor characteristics) and treatment information will be summarized descriptively. The categorical variables will be presented in the form of frequencies and percentages, while the continuous variables will be presented by mean, standard deviation and minimum and maximum values.

A logistic model will be used for the analysis of clinical benefit (categorical variable), while for the analysis of time-to-event indicators a proportional hazard model will be used. For both analyses, the optimal model will be chosen with the method of "backward" selection. A threshold value of 5% will be used to include predictive variables in the model. The estimates derived by the final models will be evaluated using a penalized model for the evaluation of maximal probability, according to the Firth approach.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* female sex
* Performance Status (ECOG) 0-2;
* hormonal-receptor positive breast cancer (Estrogen and / or Progesterone positive), HER2 negative, with evidence of stage IV / locally advanced inoperable disease
* Radiologically documented progression in 1st line treatment with Hormonal Therapy (Aromatase inhibitor / Fulvestrant) + CDK4-6i (Palbociclib / Ribociclib / Abemaciclib)
* Execution of at least one subsequent therapeutic line chosen by the clinician, with at least one radiological re-evaluation during this treatment by 31 December 2020.
* Radiologically measurable or evaluable lesions
* Written informed consent

Exclusion Criteria:

* age <18 years
* previous neoplastic pathology, within 5 years of the last active treatment
* Previous chemotherapy treatments, with biological or endocrine therapies for advanced disease, different from first-line therapy with OT + CDK4 / 6i

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the analysis of patients with HR + / HER2- advanced breast cancer treated in the second line after initial treatment failure (aromatase inhibitor or Fulvestrant + CDK4 / 6i [Palbociclib, Ribociclib or Abemaciclib]).
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Description of the choices for second line treatment in patients affected by advanced HR+/HER2- breast cancer who progressed after CDK4/6i in association with hormonal therapy. | Entire study duration, approximately 12 months
  Description of the choices for second line treatment, in the normal clinical practice of the centers adhering to the Hermione Network, in patients affected by advanced HR+/HER2- breast cancer who progressed after CDK4/6i in association with hormonal therapy.

SECONDARY OUTCOMES:
progression-free survival | from date of treatment beginning until the date of first documented progression or date of death from any cause, assessed up to 72 months
  time from the start of treatment to evidence of disease progression or death
response rate | Entire study duration, approximately 12 months
  radiological response rate according to RECIST criteria, classified as CR (Complete Response), PR (Partial Response), SD (Stable Disease), PD (Progressive Disease)
Survival Post Progression | from date of treatment beginning until the date of first documented progression or date of death from any cause, assessed up to 72 months
  survival evaluated from from date of treatment beginning until the date of first documented progression or date of death from any cause
progression by location (visceral versus non-visceral). | from date of treatment beginning until the date of first documented progression or date of death from any cause, assessed up to 72 months
  time from the date second-line treatment beginning to the date of disease progression or death from any cause, stratified according to visceral versus non-visceral diseaes
Drug toxicities | Entire study duration, approximately 12 months
  Evaluation of drug related toxicities listed according to the different therapeutic options
Physician's reasons for treatment choice in real world experience | Entire study duration, approximately 12 months
  Evaluation of the physician's reasons for treatment choice of the second-line therapy after progression to CDK4 / 6i associated with hormonal therapy
Predictive factors of response | Entire study duration, approximately 12 months
  Evaluation of predictive factors of response through the comparison of four variables according to AIC e R2 criteria

CONTACTS AND LOCATIONS:
Locations (29):
- Italy (29):
  - Clinica Oncologica Aou Ospedali Riuniti, Ancona
  - Ospedale Cardinal Massaia Asti, Asti
  - Ospedale San Martino, Belluno
  - OSPEDALE Sacro Cuore di Gesù - Fatebenefratelli, Benevento
  - Spedali Civili Brescia, Brescia
  - Ospedale Sant'Anna, San Fermo della Battaglia, Como
  - ASST Cremona - Area Donna, Cremona
  - ASST VALLE OLONA - Presidio Gallarate - SC Oncologia, Gallarate
  - A.S.S.T. Ovest Milanese, Legnano
  - Ospedale Civile di Livorno, Azienda USL Toscana Nord Ovest, Livorno
  - ISTITUTO ROMAGNOLO per la cura e lo studio dei tumori (IRST-IRCCS), Meldola
  - ASST Fatebenefratelli Sacco, Milan
  - Policlinico di Milano Ospedale Maggiore, Fondazione IRCCS Ca' Granda, Milan
  - Ospedale San Gerardo, Monza
  - UO Aziendale Olbia, Olbia
  - Ospedale La Maddalena, Palermo
  - ICS Maugeri Spa-SB PAVIA, Pavia
  - U.O.C Oncologia Ospedale "G Da Saliceto", Piacenza
  - UO Oncologia Medica I Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda USL - Arcispedale S. Maria Nuova IRCCS, Reggio Emilia
  - A.S.S.T. Rhodense Ospedale Di Circolo Rho, Rho
  - Oncologia Ospedale di Rimini, Rimini
  - IRCCS Istituto Nazionale Tumori - IFO Regina Elena, Oncologia Medica B, Roma
  - Policlinico Gemelli, Roma
  - AOU città della scienza e della salute SCDO4, Torino
  - AOU città della scienza e della salute SCDU1, Torino
  - Oncologia Trento, Trento
  - PIA FONDAZIONE Cardinale PANICO Tricase - Lecce, Tricase
  - ASST SETTELAGHI - Oncologia Varese, Varese

IPD SHARING:
Plan to Share IPD: Undecided